CLINICAL TRIAL: NCT00929383
Title: An International Registry of the Wingspan™ Stent System for the Treatment of Intracranial Atherosclerotic Stenosis
Acronym: IRISS
Status: Completed | Type: Observational
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: IRISS
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2012-09

CONDITIONS: Intracranial Atherosclerosis
Keywords: Intracranial Atherosclerosis; Stenosis; ICAD; atherosclerotic lesions; stenting
MeSH Terms: conditions — Intracranial Arteriosclerosis; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Wingspan Stent System with Gateway PTA Balloon Catheter — The Wingspan Stent System is used in conjunction with Gateway PTA Balloon Catheter to improve cerebral artery lumen diameter in patients with intracranial atherosclerotic disease.
  The Gateway Balloon Catheter is indicated for balloon dilation of the stenotic portion of intracranial arteries prior to stenting the artery for the purpose of improving intracranial perfusion.
  Other Names: Wingspan™ Stent System; 3.5F Delivery Catheter (pre-loaded with Wingspan™ Stent); Gateway™ Over-The-Wire PTA Balloon Catheter; Rotating Hemostatic Valve

SUMMARY:
The IRISS study is designed to collect clinical and angiographic outcomes data when stenting intracranial atherosclerotic lesions using the Wingspan™ Stent System with Gateway™ PTA Balloon Catheter in routine clinical practice.

DETAILED DESCRIPTION:
The Wingspan™ Stent System and Gateway™ PTA Balloon Catheter have CE mark and are commonly used in Europe. All the data collected in this registry will be from patients treated according to the physician's choice, per instructions for use, per approved indications and per local standard of care. The results from this registry will provide an understanding of the use and outcomes associated with the Wingspan™ Stent in a real world setting.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic stenosis of one of those intracranial arteries: Internal carotid artery (ICA ), M1 segment of the MCA, V4 segment of vertebral artery, basilar artery
* A Modified Rankin Score of ≤ 3
* A target vessel diameter between 2mm and ≤ 4.5mm
* Length of the target lesion of ≤ 14 mm
* Patient older than 40 years old

Exclusion Criteria:

* Patient previously stented at the target lesion
* Intracranial stenosis related to disease such as: arterial dissection, Moya Moya disease, vasculitis, radiation induced vasculopathy or fibromuscular dysplasia
* Complete occlusion of the artery on the imaging assessment
* Contraindications to antithrombotic and/or anticoagulant therapies
* Women who are pregnant or breast-feeding
* Patient not likely to be available for follow-up
* Patient protected by the law (safeguard of justice, supervision or trusteeship)

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic intracranial atherosclerotic stenosis. Patients will be included who are eligible for endovascular treatment and for which treatment with the Wingspan™ Stent system has been judged necessary by the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2009-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Houdart, Principal Investigator; Marius Hartmann, Principal Investigator
Locations (19):
- France (10):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - CHU Dijon-Hopital General, Dijon
  - CHU Limoges, Limoges
  - Höpital Gui de Chauliac, Montpellier
  - CHU Hôpital Guillaume et René Laënnec, Nantes
  - Hôpital Saint-Roch, Nice
  - Hôpital Lariboisière, Paris
  - Fondation Rotschild, Paris
  - CHU Reims, Reims
  - CHU Toulouse, Toulouse
- Germany (9):
  - Klinikum Augsburg, Augsburg
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - UKSH Campus Kiel, Kiel

REFERENCES:
- [Background] Sacco RL, Kargman DE, Gu Q, Zamanillo MC. Race-ethnicity and determinants of intracranial atherosclerotic cerebral infarction. The Northern Manhattan Stroke Study. Stroke. 1995 Jan;26(1):14-20. doi: 10.1161/01.str.26.1.14. PMID 7839388
- [Background] EC/IC Bypass Study Group. Failure of extracranial-intracranial arterial bypass to reduce the risk of ischemic stroke. Results of an international randomized trial. N Engl J Med. 1985 Nov 7;313(19):1191-200. doi: 10.1056/NEJM198511073131904. PMID 2865674
- [Background] Chimowitz MI, Lynn MJ, Howlett-Smith H, Stern BJ, Hertzberg VS, Frankel MR, Levine SR, Chaturvedi S, Kasner SE, Benesch CG, Sila CA, Jovin TG, Romano JG; Warfarin-Aspirin Symptomatic Intracranial Disease Trial Investigators. Comparison of warfarin and aspirin for symptomatic intracranial arterial stenosis. N Engl J Med. 2005 Mar 31;352(13):1305-16. doi: 10.1056/NEJMoa043033. PMID 15800226
- [Background] Kasner SE, Chimowitz MI, Lynn MJ, Howlett-Smith H, Stern BJ, Hertzberg VS, Frankel MR, Levine SR, Chaturvedi S, Benesch CG, Sila CA, Jovin TG, Romano JG, Cloft HJ; Warfarin Aspirin Symptomatic Intracranial Disease Trial Investigators. Predictors of ischemic stroke in the territory of a symptomatic intracranial arterial stenosis. Circulation. 2006 Jan 31;113(4):555-63. doi: 10.1161/CIRCULATIONAHA.105.578229. Epub 2006 Jan 23. PMID 16432056
- [Background] Connors JJ 3rd, Wojak JC. Percutaneous transluminal angioplasty for intracranial atherosclerotic lesions: evolution of technique and short-term results. J Neurosurg. 1999 Sep;91(3):415-23. doi: 10.3171/jns.1999.91.3.0415. PMID 10470816
- [Background] Marks MP, Wojak JC, Al-Ali F, Jayaraman M, Marcellus ML, Connors JJ, Do HM. Angioplasty for symptomatic intracranial stenosis: clinical outcome. Stroke. 2006 Apr;37(4):1016-20. doi: 10.1161/01.STR.0000206142.03677.c2. Epub 2006 Feb 23. PMID 16497979
- [Background] SSYLVIA Study Investigators. Stenting of Symptomatic Atherosclerotic Lesions in the Vertebral or Intracranial Arteries (SSYLVIA): study results. Stroke. 2004 Jun;35(6):1388-92. doi: 10.1161/01.STR.0000128708.86762.d6. Epub 2004 Apr 22. PMID 15105508
- [Background] Wojak JC, Dunlap DC, Hargrave KR, DeAlvare LA, Culbertson HS, Connors JJ 3rd. Intracranial angioplasty and stenting: long-term results from a single center. AJNR Am J Neuroradiol. 2006 Oct;27(9):1882-92. PMID 17032860
- [Background] Bose A, Hartmann M, Henkes H, Liu HM, Teng MM, Szikora I, Berlis A, Reul J, Yu SC, Forsting M, Lui M, Lim W, Sit SP. A novel, self-expanding, nitinol stent in medically refractory intracranial atherosclerotic stenoses: the Wingspan study. Stroke. 2007 May;38(5):1531-7. doi: 10.1161/STROKEAHA.106.477711. Epub 2007 Mar 29. PMID 17395864
- [Background] Levy EI, Turk AS, Albuquerque FC, Niemann DB, Aagaard-Kienitz B, Pride L, Purdy P, Welch B, Woo H, Rasmussen PA, Hopkins LN, Masaryk TJ, McDougall CG, Fiorella DJ. Wingspan in-stent restenosis and thrombosis: incidence, clinical presentation, and management. Neurosurgery. 2007 Sep;61(3):644-50; discussion 650-1. doi: 10.1227/01.NEU.0000290914.24976.83. PMID 17881980
- [Background] Zaidat OO, Klucznik R, Alexander MJ, Chaloupka J, Lutsep H, Barnwell S, Mawad M, Lane B, Lynn MJ, Chimowitz M; NIH Multi-center Wingspan Intracranial Stent Registry Study Group. The NIH registry on use of the Wingspan stent for symptomatic 70-99% intracranial arterial stenosis. Neurology. 2008 Apr 22;70(17):1518-24. doi: 10.1212/01.wnl.0000306308.08229.a3. Epub 2008 Jan 30. PMID 18235078
- [Background] Fiorella D, Woo HH. Emerging endovascular therapies for symptomatic intracranial atherosclerotic disease. Stroke. 2007 Aug;38(8):2391-6. doi: 10.1161/STROKEAHA.107.482752. Epub 2007 Jun 21. No abstract available. PMID 17585085
- [Background] Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) Trial Investigators. Design, progress and challenges of a double-blind trial of warfarin versus aspirin for symptomatic intracranial arterial stenosis. Neuroepidemiology. 2003 Mar-Apr;22(2):106-17. doi: 10.1159/000068744. No abstract available. PMID 12656117
- [Background] Samuels OB, Joseph GJ, Lynn MJ, Smith HA, Chimowitz MI. A standardized method for measuring intracranial arterial stenosis. AJNR Am J Neuroradiol. 2000 Apr;21(4):643-6. PMID 10782772

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients eligible were diagnosed with symptomatic Intracranial Atheroslcerotic disease and scheduled to be treated with a Wingspan Stent in 6 centers in France and 9 centers in Germany.
  The first patient was enrolled on 11 March 2009 and last patient on 30 April 2012.
Pre-assignment Details: This was an open label registry (observational study). All patients scheduled for treatment with a Wingspan Stent meeting inclusion/exclusion criteria were eligible for participation.
Groups:
- Wingspan: Prospective, open label study of patients with symptomatic Intracranial Atherosclerotic disease scheduled for treatment with the Wingspan Stent and Gateway balloon system. The patients were treated endovascularly as per standard of care at each study site
Period: Overall Study
Arm/Group | Wingspan
Started | 82
Completed | 67
Not Completed | 15

BASELINE CHARACTERISTICS:
Population: Prospective, open label registry. All patients meeting inclusion/exclusion at the study centers were eligible for paritcipation.
  As this was an observational registry, no statistical hypothesis was stated a priori.
Groups:
- Patients Treated With a Wingspan Stent: Prospective, single arm, open label study of patients with symptomatic Intracranial Atherosclerotic disease scheduled for treatment with the Wingspan Stent and Gateway balloon system. The patients were treated endovascularly as per standard of care at each study site
Arm/Group | Patients Treated With a Wingspan Stent
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.23 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 60

OUTCOME MEASURES:

1. Primary Outcome: Successful Wingspan™ Stent Implantation (Access to the Lesion With the Stent, Accurate Deployment of the Stent Across the Target Lesion)
Description: The number of Wingspan Stents successfully deployed across the target lesion.
Time Frame: Peri-procedural
Population: (ITT) Intent-to-treat
Measure: Number; unit: patients w stent implanted
Groups:
- Patients Treated With a Wingspan Stent: Prospective, open label study of patients with symptomatic Intracranial Atherosclerotic disease scheduled for treatment with the Wingspan Stent and Gateway balloon system. The patients were treated endovascularly as per standard of care at each study site
Arm/Group | Patients Treated With a Wingspan Stent
Number analyzed (Participants) | 82
patients w stent implanted | 78

2. Primary Outcome: Cumulative Morbidity and Mortality Rate (Ischemic Event, Parenchymal Brain Hemorrhage, Subarachnoid or Intraventricular Hemorrhage or Death)
Description: Any stroke or neurological death at </= 30 days will be included in the cumulative morbidity and mortality rate.
  There was a 14.6% rate of cumulative morbidity and mortality at 30 days comprised of 12 events/82 patients.
Time Frame: 30 days
Population: (ITT) Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Patients Treated With a Wingspan Stent
Number analyzed (Participants) | 82
participants | 12

3. Primary Outcome: Rate of Recurrent Ischemic Stroke in the Target Territory
Description: The rate of recurrent ischemic stroke from 31 days to 12 months post procedure was 1.3% or 1 event per 77 patients analyzed.
Time Frame: 12 Months
Population: (ITT) Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Patients Treated With a Wingspan Stent
Number analyzed (Participants) | 77
participants | 1

4. Secondary Outcome: Cumulative Stroke Rate at 12 Months
Description: The cumulative stroke rate at 12 months (any stroke or neurological death </= 30 days or any ischemic stroke in territory >/= 31 days is 15.9% or 13 events per 82 patients
Time Frame: 12 months
Population: (ITT) Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Patients Treated With a Wingspan Stent
Number analyzed (Participants) | 82
participants | 13

5. Secondary Outcome: Rate of Restenosis
Description: The rate of restenosis at 12 months was defined as the degree of residual stenosis greater than 50% as determined by the study sites using the WASID method. There was a 10.4% rate of restenosis >50% or 8 patients out of 77 analyzed. The differences in this analysis population N=77 vs. ITT N= 82 populations results from exclusion of N=4 patients with no stent implanted and N=1 patient who died prior to any follow up measures of restenosis.
  The WASID method is a standardized protocol for measuring intracranial arterial stenosis.
  [1-(Dstenosis/Dnormal)] x100=% stenosis (where D=vessel diameter)
Time Frame: 12 Months
Population: There were only N=77 patients available for analysis of restenosis at 12 months. This differs from the original N=82 ITT population in that denominator is based on the number of subjects available at 30 day follow up. Five subjects who exited the study at discharge were excluded from the analysis (no stent implanted (4), death (1)).
Measure: Number; unit: participants
Arm/Group | Patients Treated With a Wingspan Stent
Number analyzed (Participants) | 77
participants | 8

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the procedure until last follow up visit (12 months).
Description: Serious Adverse Events include adverse events that result in death, require either inpatient hospitalization or the prolongation of hospitalization, are life-threatening, result in a persistent or significant disability/incapacity or result in a congenital anomaly/birth defect.
Arm/Group | Wingspan
Serious Adverse Events (participants affected / at risk) | 29/82
Other Adverse Events (participants affected / at risk) | 5/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wingspan (N=82)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Catheter site hematoma (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 4 (4)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 12 (12)
Convulsion (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Neurological decompensation (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 5 (6)
Renal cancer (Renal and urinary disorders) | 1 (1)
Urethral cancer (Renal and urinary disorders) | 1 (1)
Artery dissection (Vascular disorders) | 1 (1)
Thrombosis in device (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wingspan (N=82)
Conjunctivitis (Eye disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Artery dissection (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No